CLINICAL TRIAL: NCT05693597
Title: Evaluation of the Effect of Nigella Sativa for the Prophylaxis to Radiation Induced Dermatitis in Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: German University in Cairo (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mayar Waleed Salaheldin Aly, Clinical Pharmacy Lecturer Assistant, German University in Cairo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: N.sativavsRID BreastCancerpt.
Record Dates: First submitted 2023-01-04; First posted 2023-01-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Radiation Dermatitis
Keywords: Nigella sativa; Black seed; Baraka; Radiation induced dermatitis; Breast cancer
MeSH Terms: conditions — Radiodermatitis; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Group I (control): Patients will not receive any prophylactic intervention, as there is no standard of care for prophylaxis to the radiation induced dermatitis (RID).
  Group II (Topical intervention): Patients will receive Imtenan ® N. sativa oil apply 1.5 mls; twice daily; not sooner than 2 hours before and after radiation therapy; from day 1 of radiation therapy till the end.
  Group III (Oral intervention): Patients will receive Baraka ® N. sativa gelatin capsules; 40mg/Kg/day; from day 1 of radiation therapy till the end
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (control) (No Intervention): Patients will not receive any prophylactic intervention, as there is no standard of care for prophylaxis to the radiation induced dermatitis (RID).
- Group II (Topical intervention) (Experimental): Patients will receive Imtenan ® N. sativa oil apply 1.5 mls; twice daily; not sooner than 2 hours before and after radiation therapy; from day 1 of radiation therapy till the end.
  Interventions: Drug: Imtenan Oil
- Group III (Oral intervention) (Experimental): Patients will receive Baraka ® N. sativa gelatin capsules; 40-80 mg/Kg/day; from day 1 of radiation therapy till the end
  Interventions: Drug: Baraka Capsules

INTERVENTIONS:
Drug: Imtenan Oil — Cold Press Oil
  Arms: Group II (Topical intervention)
Drug: Baraka Capsules — Soft Gelatin Capsules
  Arms: Group III (Oral intervention)

SUMMARY:
Radiation induced dermatitis (RID) is one of the leading adverse events of radiation therapy, and if occurred could alter the course of therapy. The main pathways of RID is inflammation and oxidative stress on local and systemic bases. Nigella sativa is an herbal medicine whose anti-inflammatory and antioxidant activities have been proven in several clinical trials. Thus, the aim of the present study is to evaluate the efficacy of Nigella sativa as a prophylactic method against the development of RID.

DETAILED DESCRIPTION:
Radiation induced dermatitis (RID) is one of the most commonly reported adverse events of breast radiation therapy (RT).Radiation therapy toxicity is exhibited within hours to weeks of exposure and persisting throughout the course of treatment. Radiation induced dermatitis is a result of generation of reactive oxygen species (ROSs), which in return induces epidermal and dermal inflammatory responses. Radiation causes structural tissue damage, which trigger production of pro-inflammatory mediators; as NF-κB, iNOS, COX-2, EGFR, MCP-1, and cytokines such as IL-1, IL-2, IL-6, TNF-a, and IFN- γ, and immune-stimulatory response; involving an increased movement of leukocytes from the blood into the irradiated tissues. Subsequently erythema, ulceration, and edema are developed. This is then followed by thinning of the epidermis, accompanied with degeneration of glands, which manifests as dry desquamation. If damage to the basal cells and glands is more severe, moist desquamation occur. From previous, it can be deduced that inflammatory response plays a significant role in the radiotherapy induced dermatitis.

There are many agents that are used in the management of RID in the clinical settings, however, up till now there is none supported by the guidelines. Radiation induced dermatitis occurrence, not only could it impair the patient's quality of life but it could also affect the RT course of treatment, which could negatively influence the cancer treatment. Therefore more effort is needed to find a method of prevention of RID, resulting from breast RT, especially that there is no standard of care for prophylaxis to the radiation induced dermatitis (RID).

Nigella sativa is herbal medicine that has been widely used in different parts of the world by different cultures. It has been used traditionally as a remedy for several diseases including fever, cough, chronic headache, dizziness, back pain, dysmenorrhea, obesity, diabetes, infection and inflammation, hypertension, and gastrointestinal disorders such as flatulence, and dysentery. Preclinical and clinical studies have demonstrated the anti-inflammatory, immunomodulatory, antioxidant, analgesic, and antimicrobial properties of N. sativa.

Thymoquinone (TQ) is the prominent constituent of Nigella sativa, to which the biological properties have been attributed. Thymoquinone can act as a potent free radical and superoxide radical scavenger at both nanomolar and micromolar range, respectively. As well as, its beneficial effects on antioxidant enzymes, and its detrimental effects on pro-inflammatory mediators/cytokines, and pro-inflammatory transcription factor; nuclear factor kappa B (NF-κB).

Based on literature, Nigella sativa has been shown to have antioxidant and anti-inflammatory effects. As, both the fixed oil of N. sativa, as well as thymoquinone (the main compound of the essential oil), were proven to inhibit non-enzymatic lipid peroxidation and have an appreciable free radical scavenging properties. Furthermore, orally administered Nigella sativa oil showed a reduction of IL-4 and NO production in rats. Additionally, Thymoquinone showed anti-inflammatory activity through inhibition of cyclooxygenase (COX) and 5-lipooxygenase (5-LPO), as well as through lowering TNF-α and IL-1β levels in arthritis in rats. It is worth mentioning that thymoquinone was proven to significantly reduce pancreatic ductal adenocarcinoma cell synthesis of MCP-1, TNF-a, IL-1β and Cox-2. It also inhibited the constitutive and TNF-a-mediated activation of NF-kB.

Hence, many clinical trials have been using Nigella sativa, to see its anti-inflammatory and antioxidant effects in different indications including its anti-inflammatory effect in treatment of oral mucositis in head and neck cancers patients, and managing dermatitis in breast cancer patients, and its antioxidant effect in patients with psoriasis, and acute tonsillo-pharyngitis, and many more, where Nigella sativa showed to be not only safe but effective as well. Nigella sativa oil, Baraka ® gelatin capsules, has been used in doses up to 80 mg/kg/day in children with acute lymphoblastic leukemia, in the protection against doxorubicin-induced cardiac toxicity and in the protection against Methotrexate induced hepatotoxicity, where it was effective and safe.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive, early stage breast carcinoma scheduled for adjuvant radiotherapy.
* Women aged ≥18 years.

Exclusion Criteria:

* Prior exposure to radiotherapy
* Patients with generalized skin disorder
* Patients who failed to sign the written consent

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Incidence of development of radiation induced dermatitis | 6 weeks
  If the patient developed Radiation induced dermatitis or not

SECONDARY OUTCOMES:
Evaluation of Severity of RID developed | 6 weeks
  The severity of moist desquamation assessed by Common Terminology Criteria for Adverse Events (CTCAE, version6) criteria based on the clinical presentation.
Evaluation of Pain Intensity | 6 weeks
  Pain related assessment will be done through a Visual Analog Scale, with 0 being No pain and 10 being unbearable pain
Evaluation of Incidence of Treatment-Emergent Adverse Events | 6 weeks
  Patients will be educated and instructed to report any adverse events
Evaluation of Quality of life | 6 weeks
  Skin-related quality of life assessed through the Dermatology Life Quality Index (DLQI)
Evaluation of Time to develop grade 2 RID | 6 weeks
  Time to develop grade 2 RID incidence, will be assessed by Common Terminology Criteria for Adverse Events (CTCAE, version6) criteria based on the clinical presentation.

CONTACTS AND LOCATIONS:
Overall Officials: Mayar Waleed Salaheldin Aly, M.Sc., Principal Investigator — German University in Cairo
Locations (1):
- Ain Shams University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Radiation-induced skin reactions: mechanism and treatment — https://www.dovepress.com/radiation-induced-skin-reactions-mechanism-and-treatment-peer-reviewed-fulltext-article-CMAR
- See also: Clinical practice guidelines for the prevention and treatment of acute and late radiation reactions from the MASCC Skin Toxicity Study Group — https://link.springer.com/article/10.1007/s00520-013-1896-2
- See also: The prevention and management of acute skin reactions related to radiation therapy: a systematic review and practice guideline — https://link.springer.com/article/10.1007/s00520-006-0063-4
- See also: Symptom Management Guidelines: RADIATION DERMATITIS — http://www.bccancer.bc.ca/nursing-site/Documents/Symptom%20Management%20Guidelines/14RadiationDermatitis.pdf
- See also: A Review of Medicinal Uses and Pharmacological Activities of Nigella sativa — https://scialert.net/abstract/?doi=pjbs.2004.441.451
- See also: Antioxidant activity of Nigella sativa essential oil — https://pubmed.ncbi.nlm.nih.gov/10925395/
- See also: Ameliorating effects of Nigella sativa oil on aggravation of inflammation, oxidative stress and cytotoxicity induced by smokeless tobacco extract in an allergic asthma model in Wistar rats — https://pesquisa.bvsalud.org/portal/resource/pt/ibc-177883
- See also: Anti-Inflammatory Effect of Nigella Sativa Oil on Chemoradiation-Induced Oral Mucositis in Patients With Head and Neck Cancers — https://innovareacademics.in/journals/index.php/ijcpr/article/view/35704
- See also: Evaluation of efficacy, safety and antioxidant effect of Nigella sativa in patients with psoriasis: A randomized clinical trial — https://www.jceionline.org/article/evaluation-of-efficacy-safety-and-antioxidant-effect-of-nigella-sativa-in-patients-with-psoriasis-a-3557
- See also: Symptomatic treatment of acute tonsillo-pharyngitis patients with a combination of Nigella sativa and Phyllanthus niruri extract — https://www.dustri.com/article_response_page.html?artId=4697&doi=10.5414/CPP46295&L=0
- See also: Protective role of black seed oil in doxorubicin-induced cardiac toxicity in children with acute lymphoblastic leukemia — https://europepmc.org/article/med/31964219
- See also: Protective Effect of Nigella sativa Oil against Methotrexate Induced Hepatotoxicity in Children with Acute Lymphoblastic Leukemia — https://www.longdom.org/open-access/protective-effect-of-nigella-sativa-oil-against-methotrexate-induced-hepatotoxicity-in-children-with-acute-lymphoblastic-leukemia-2329-6917.1000123.pdf
- See also: Effectiveness of Nigella sativa Oil in the Management of Rheumatoid Arthritis Patients: A Placebo Controlled Study — https://tahomaclinic.com/Private/Articles3/RA/Gheita%202012%20-%20Effectiveness%20of%20Nigella%20sativa%20oil%20in%20rheumatoid%20arthritis.pdf
- See also: Effect of Nigella sativa (black seed) on subjective feeling in patients with allergic diseases — https://pubmed.ncbi.nlm.nih.gov/14669258/
- See also: Dermatology Life Quality Index (DLQI)-a simple practical measure for routine clinical use — https://europepmc.org/article/med/8033378